CLINICAL TRIAL: NCT00637351
Title: A Study to Collect Blood and Urine Samples in Elderly Subjects With Pneumonia to Support the Development of Bacteriological Diagnostic Assays
Brief Title: A Study in Elderly Subjects With Pneumonia to Support the Development of Bacteriological Diagnostic Assays
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111074
Record Dates: First submitted 2008-03-10; First posted 2008-03-18 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Infections, Streptococcal
MeSH Terms: conditions — Streptococcal Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, urine samples

GROUPS / COHORTS (2):
- Group A: Subjects with diagnosed pneumonia & positive culture of streptococcus pneumoniae
  Interventions: Procedure: Blood sample; Procedure: Urine sample
- Group B: Subjects with diagnosed pneumonia & positive culture of non-typable haemophilus influenzae
  Interventions: Procedure: Blood sample; Procedure: Urine sample

INTERVENTIONS:
Procedure: Blood sample — One blood sample will be collected at the time of screening for subjects
Procedure: Urine sample — One urine sample will be collected at the time of screening for subjects

SUMMARY:
GSK Biologicals is working on the development of a vaccine to protect elderly people from bacterial pneumonia. Diagnostic of bacterial pneumonia is difficult, and for the future studies in that project, it would be useful to have some easy non invasive tests. New clinical read-outs are needed to detect and identify the causative pathogen. These assays will be based on specific antigen detection in the urine or specific pathogen DNA detection in the blood. Technical and clinical validation of these assays will be realised at later stage with samples coming from epidemiological and/or phase III studies.

To allow the development of such tests in GSK Biologicals laboratories, urine and blood samples are needed from subjects aged 65 or above who have diagnosed pneumonia.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female aged 65 or above at the time of the study.
* Written informed consent obtained from the subject.
* Clinical pneumonia diagnosed by chest X-ray detected within 7 days before study entry.

Exclusion Criteria:

* Vaccination with a pneumococcal or Haemophilus vaccine within the last 3 months before study entry.
* Antibiotherapy started more than 7 days before Screening.
* A negative culture for Streptococcus pneumoniae or Non-Typable Haemophilus influenza.
* A urine sample at Screening less than 40 mL.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly subjects with diagnosed pneumonia
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2008-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Detection of Streptococcus pneumoniae antigens in the urine of subjects with diagnosed pneumonia. | At the time of analysis.
Detection of Streptococcus pneumoniae DNA in the blood of subjects with diagnosed pneumonia. | At the time of analysis.

SECONDARY OUTCOMES:
Detection of Non-Typable Haemophilus influenzae antigens in the urine of subjects with diagnosed pneumonia. | At the time of analysis.
Detection of Non-Typable Haemophilus influenzae DNA in the blood of subjects with diagnosed pneumonia. | At the time of analysis.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Yvoir